CLINICAL TRIAL: NCT00596804
Title: A Phase I Study of Immunotherapy With hA20 Administered Once Weekly for 4 Consecutive Weeks in Patients With CD20+ Non- Hodgkin's Lymphoma
Brief Title: Safety Study of Different Doses of hA20 (Veltuzumab) in CD20+ Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hA20-01EU
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2012-02

CONDITIONS: Non-Hodgkin's Lymphoma; Lymphoma, Diffuse; Lymphoma, Diffuse, Mixed Lymphocytic-Histiocytic
Keywords: NHL; Non-Hodgkin's lymphoma; follicular lymphoma; B-cell lymphoma; diffuse large cell lymphoma; small lymphoctytic lymphoma; Mantle cell lymphoma; MALT; marginal zone lymphoma; High-Grade; Intermediate-Grade; Low-Grade; Mixed
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — veltuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: veltuzumab — once weekly intravenous dosing for 4 weeks
  Other Names: IMMU-106; hA20; humanized anti-CD20

SUMMARY:
This study is being done to assess the safety and tolerance of different doses of humanized hA20 in patients with NHL.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years old
* Histological diagnosis of CD20+ B-cell NHL (all grades) by WHO lymphoma criteria
* Failed at least one prior standard chemotherapy regimen for NHL
* Failed rituximab treatment for relapsed NHL
* Measurable NHL disease by CT, with at least one lesion >1.5 cm in one dimension
* Adequate performance status (>70 Karnofsky scale, 0-1 ECOG) with an estimated life expectancy of at least 6 months
* Adequate hematologic status, without ongoing transfusional support (hemoglobin ≥ 10 g/dL, ANC ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L)
* Adequate renal and hepatic function, defined as: creatinine ≤ 1.5 x Institution Upper Limit of Normal (IULN), bilirubin ≤ 1.5 x IULN, AST and ALT ≤ 2.5 x IULN
* Otherwise, <Grade 1 toxicity at study entry by NCI CTC version 2.0, including recovery from all acute toxicities incurred as a result of previous surgery, radiotherapy or chemotherapy, whether investigational or conventional.
* At least 6 months beyond previous rituximab treatment, 12 weeks beyond autologous stem cell transplant, 4 weeks beyond chemotherapy, other experimental treatments, or any radiation therapy to the index lesion(s).
* Ability to provide signed, informed consent

Exclusion Criteria:

* Pregnant or lactating women. Women of childbearing potential are required to have a negative pregnancy test
* Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control while enrolled in the study until at least 12 weeks after the last weekly hA20 infusion.
* Rituximab resistant, defined as having progressed during or within 6 months of rituximab treatment.
* Excessive toxicity to rituximab (NCI CTC Grade 3 or 4) or known to be HACA positive
* Prior radioimmunotherapy, including Zevalin or Bexxar,
* Prior therapy with other human or humanized monoclonal antibodies, unless HAHA tested and negative
* Primary CNS lymphoma, HIV lymphoma or transformed lymphoma, or presence of symptomatic CNS metastases or carcinomatous meningitis.
* Bulky disease by CT, defined as any single mass >10 cm in its greatest diameter
* Pleural effusion with positive cytology for lymphoma Known to be HIV positive, or hepatitis B or C positive
* Known autoimmune disease or presence of autoimmune phenomena.
* Evidence of infection or requiring antibiotics within 5 days.
* Corticosteroid use within 2 weeks
* Prior malignancy with less than a 5-year disease-free interval, excluding nonmelanoma skin cancers and carcinoma in situ of the cervix.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of studyprocedures and follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety of hA20 with this administration schedule and dosing | first 12 weeks, then over 2 years
tolerance of hA20 with this administration schedule and dosing | first 12 weeks
immunogenicity of hA20 with this administration schedule and dosing | first 12 weeks, as needed over 2 years

SECONDARY OUTCOMES:
Pharmacodynamics of hA20 | first 12 weeks, then up to 2 years
pharmacokinetics hA20 | first 12 weeks, then up to 2 years
assess efficacy | 4 and 12 weeks, then every 3 months for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (3):
- France (2):
  - Service Des Maladies Du Sang, Lille, Cedex
  - Centre hospitalier Lyon, Lyon, Pierre Benite Cedex
- University of Leicester, Leicester, United Kingdom

REFERENCES:
- [Background] Stein R, Qu Z, Chen S, Rosario A, Shi V, Hayes M, Horak ID, Hansen HJ, Goldenberg DM. Characterization of a new humanized anti-CD20 monoclonal antibody, IMMU-106, and Its use in combination with the humanized anti-CD22 antibody, epratuzumab, for the therapy of non-Hodgkin's lymphoma. Clin Cancer Res. 2004 Apr 15;10(8):2868-78. doi: 10.1158/1078-0432.ccr-03-0493. PMID 15102696
- [Background] Stein R, Qu Z, Chen S, Solis D, Hansen HJ, Goldenberg DM. Characterization of a humanized IgG4 anti-HLA-DR monoclonal antibody that lacks effector cell functions but retains direct antilymphoma activity and increases the potency of rituximab. Blood. 2006 Oct 15;108(8):2736-44. doi: 10.1182/blood-2006-04-017921. Epub 2006 Jun 15. PMID 16778139
- [Background] Goldenberg DM, Morschhauser F, Wegener WA. Veltuzumab (humanized anti-CD20 monoclonal antibody): characterization, current clinical results, and future prospects. Leuk Lymphoma. 2010 May;51(5):747-55. doi: 10.3109/10428191003672123. PMID 20214444
- [Result] Franck Morschhauser1*, John P Leonard2, Bertrand Coiffier3*, et.al. INITIAL SAFETY AND EFFICACY RESULTS OF A SECOND-GENERATION HUMANIZED ANTI-CD20 ANTIBODY, IMMU-106 (HA20), IN NON-HODGKINS LYMPHOMA: ASH abstract 2005.
- [Result] Morschhauser F, Leonard JP, Coiffier B Petillon M, Coleman M,. Bahkti A, Teoh N, Wegener WA, Goldenberg DM. Phase I/II result of a seoncd-generation humanized anti- CD20 antibody, IMMU-106 (.hA20), in NHL: 2006 ASCO Annual Meeting.Proceedings; 24/18S Part I of II:429s
- [Result] Morschhauser F, Leonard JP, Fayad L, Coiffier B, Petillon M, Coleman M,. Horne H, Teoh N, Wegener WA, Goldenberg DM. Low doses of humanized anti-CD20 antibody, IMMU-106 (hA20), in refractory or recurrent NHL: Phase I/II results. 2007 ASCO Annual Meeting.Proceedings; 25/18S Part I of II:449s
- [Result] Morschhauser F, Leonard JP, Fayad L, Coiffier B, Petillon MO, Coleman M, Schuster SJ, Dyer MJ, Horne H, Teoh N, Wegener WA, Goldenberg DM. Humanized anti-CD20 antibody, veltuzumab, in refractory/recurrent non-Hodgkin's lymphoma: phase I/II results. J Clin Oncol. 2009 Jul 10;27(20):3346-53. doi: 10.1200/JCO.2008.19.9117. Epub 2009 May 18. PMID 19451441